CLINICAL TRIAL: NCT05798312
Title: Randomized and Multicenter Study to Evaluate the Impact of a Customizable Support Material in the Knowledge and Satisfaction of Breast Cancer Patients
Brief Title: Randomized and Multicenter Study to Evaluate a Customizable Support Breast Cancer Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicos e Investigadores en la Lucha contra el Cancer de Mama (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Cynthia Villarreal Garza, MD, DSc, Medicos e Investigadores en la Lucha contra el Cancer de Mama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IMAP-CM
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Knowledge, Attitudes, Practice; Patient Empowerment; Patient Satisfaction
Keywords: breast cancer; patient education; written information; shared decision making; Latin America
MeSH Terms: conditions — Breast Neoplasms; Behavior; Patient Participation; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The intervention group will receive customizable support material while the standard group will receive a non-customizable material.
Who Masked: Participant
Masking Description: Paticipants will receive a support material with information about breast cancer. Those in the intervention group will not know of the existence of a non-customizable material and those in the standard group will not know of the existence of a customizable material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive customizable support material.
  Interventions: Other: Customizable support material
- Standard group (Sham Comparator): The standard group will receive a non-customizable support material.
  Interventions: Other: Non-customizable support material

INTERVENTIONS:
Other: Customizable support material — Customizable support material will enable patients to identify their personal breast cancer information.
  Arms: Intervention group
Other: Non-customizable support material — Non-customizable support material will include general breast cancer information.
  Arms: Standard group

SUMMARY:
The goal of this clinical trial is to evaluate if a customizable support material allows to improve the knowledge about the stage and subtype of the disease, as well as the indicated treatments, in comparison with a non-customizable support material among patients with breast cancer.

The main question it aims to answer is:

• What is the impact of delivering a customizable support material so that patients with breast cancer know and remember the stage and subtype of their disease, as well as the indicated treatments, compared to non-customizable support material?

Participants in the intervention group will be provided customizable support material while those in the standard group will receive a non-customizable material.

DETAILED DESCRIPTION:
In the present investigation, it is planned to carry out a prospective, multicenter study, randomized and blinded to the statistician. Patients with a recent diagnosis of CM and who are scheduled to have their first consultation in which their options will be discussed of treatment to participate in the study. To those who agree to participate and sign the informed consent, the protocol coordinator of each center will randomly assign them to the intervention group or the standard group (in a 1:1 ratio) before the appointment medical. The intervention group will receive customizable support material while the Standard group will receive a non-customizable material (Annex 2). Additionally, you will be instructed to the intervention group that the support material received can be filled with the information discussed with the medical team. The protocol coordinator will obtain sociodemographic data and clinicopathology of the medical records of the participants. After the next visit follow-up, the coordinator will apply to both groups questionnaires about the knowledge of the patient about his own disease, satisfaction with the support material received and perceived ability to participate in discussions about their treatment, and the comprehension of written materials (CHLT-6). After one month, both groups will respond knowledge questionnaires to assess long-term information retention, disease uncertainty (SF-MUIS) and satisfaction with medical information provided (EORTC-QLQ-INFO25).

ELIGIBILITY:
Inclusion Criteria:

* Women with a recent diagnosis of primary breast cancer treated at the participant centers
* Women who will receive information about their options for the first time treatment
* Provision of informed consent to participate in the study

Exclusion Criteria:

* Patients who have already started systemic treatment for breast cancer
* Patients with medical records not available for data collection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Knowledge | 1-month
  Evaluate if a customizable support material allows to improve the knowledge about the stage and subtype of the disease, as well as the indicated treatments, in comparison with a non-customizable support material as measured by the knowledge questionnaire assessing patients' knowledge of their disease extension (in situ vs invasive cancer); clinical stage; estrogen, progesterone and HER2 receptor status; and treatments to which they are candidates.

SECONDARY OUTCOMES:
Patient satisfaction | 1-month
  Assess patient satisfaction with the written information provided and the perception of their ability to actively participate in discussions about the treatment when offered a customizable educational brochure and compare it to the patients receiving a non-customizable brochure
Comprehension | 1-month
  Determine if the comprehension of written materials (customizable or not customizable) is associated with the level of health literacy (Health Literacy) as measured by the Cancer Health Literacy Test - 6 (CHLT-6) instrument
Satisfaction with medical information | 1-month
  To determine if satisfaction with medical information is higher when offered a customizable vs. non-customizable educational brochure as per measured by the European Organization for Research and Treatment of Cancer test Quality of Life Group information questionnaire (EORTC QLQ-INFO 25)
Illness uncertainty | 1-month
  Determine if the uncertainty of the disease with the medical information is lower when offered a customizable educational brochure versus offering non-customizable material, as measured by the short form of Mishel Uncertainty Illness Scale (SF-MUIS)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Zambrano Hellion, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villarreal-Garza C, Ferrigno AS, De la Garza-Ramos C, Vazquez-Juarez D, Moreno-Jaime B, Remolina-Bonilla Y, Segura-Gonzalez M, Mariscal-Ramirez I, Perazzo F, Garnica-Jaliffe G, Neciosup-Delgado S, Conde-Flores E, Mysler S, Hernandez-Ayala A, Barajas-Sanchez A, Rios Mercado MDS, Noh-Vazquez NM, Garcia-Rodriguez R, Platas A, Tamez-Salazar J, Mireles-Aguilar T, Platas A. Effect of receiving a customizable brochure on breast cancer patients' knowledge about their diagnosis and treatment: A randomized clinical trial. Cancer Med. 2023 Jul;12(14):15612-15627. doi: 10.1002/cam4.6215. Epub 2023 Jun 14. PMID 37317676